CLINICAL TRIAL: NCT04600310
Title: A Randomized, Single-blinded Trial to Study the Efficacy, Safety, and Time Saving Using the ULTRAPREP Device With FDA Approved Antisepsis Solution (70% Isopropyl Alcohol and 2% Chlorhexidine) in Preoperative Skin Antisepsis.
Brief Title: ULTRAPREP Used to Perform Skin Antisepsis Outside the Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prep Tech, LLC (Other)
Responsible Party: Principal Investigator, Mallory M. Przybylski, DPM, MSc, Principal Investigator, Prep Tech, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ULTRAPREP-100
Record Dates: First submitted 2020-09-29; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Time Saved Performing Skin Antisepsis Process Outside the OR; Antisepsis of Skin Preparation Outside the OR
Keywords: skin antisepsis; OR efficiency

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study Arm 1 Conventional Prep/Control (Other): The preoperative preparation for the control group will use ChloraPrep (2% chlorhexidine and 70% isopropyl alcohol) that will be applied to the skin using a sponge-on-a-stick method; this solution is widely recognized as optimal. After the alcohol-based solution has evaporated (no less than 3 minutes), the patient extremity is draped for surgery.
  Interventions: Device: No Intervention
- Study Arm 2 ULTRAPREP Group/Intervention Arm (Other): ChloraPrep (2% chlorhexidine and 70% isopropyl alcohol) will be poured into the ULTRAPREP bag which will be placed on the patient's extremity while in the holding area; it will be removed only after scrub time of 3 minutes is complete and the patient has been transferred to the OR, anesthetized, and positioned. The patient is draped only after the solution has evaporated (no less than 3 minutes).
  Interventions: Device: ULTRAPREP

INTERVENTIONS:
Device: ULTRAPREP — ULTRAPREP device for reducing OR prep times.
  Arms: Study Arm 2 ULTRAPREP Group/Intervention Arm
Device: No Intervention — Conventional skin preparation technique
  Arms: Study Arm 1 Conventional Prep/Control

SUMMARY:
Testing ULTRAPREP (consists of a clear bag sealed on one end with the other end enclosing the patients extremity) for safety and efficacy to perform skin antisepsis outside the operating room.

DETAILED DESCRIPTION:
The purpose of the study is to determine if ULTRAPREP is equal to or better than the conventional methods of preoperative skin antisepsis (the technique of cleansing the skin to help prevent infection) in surgical cases. The study will also help determine if ULTRAPREP will decrease the total amount of time in the operating room. The study will focus on whether or not using ULTRAPREP provides better patient flow and patient safety while improving a surgical staff's workload and workflow. The study includes 2 study arms:

Study Arm #1: the conventional method (or standard of care) will use an accepted skin disinfectant solution with ChloraPrep (70% isopropyl alcohol and 2% chlorhexidine). The solution is "painted" on the patient's skin using a sponge on a stick. The application time is with this method is 3 minutes plus 3 minutes for solution to evaporate. This is a widely-accepted method used in ORs. The preparation process is performed by surgical staff in the OR prior to surgery.

Study Arm #2: using ULTRAPREP bag containing ChloraPrep (70% isopropyl alcohol and 2% chlorhexidine). The bag will be placed on the patient's lower extremity in the holding area. The lower extremity will be scrubbed for 3 minutes. Once the patient is transferred to the OR, the solution will be suctioned out of the bag and the bag removed from the lower extremity to allow the solution to evaporate, this process take 3 minutes. the patient is then draped for surgery.

This study consists of 57 patients in each arm.

Sterile culture swabs will be taken from toenail beds and between toes or from fingernail beds and between fingers, depending on surgery site. The cultures will be taken preoperative before any disinfecting has begun and just before patient extremity is draped (after allowing 3 minutes for alcohol in disinfectant to evaporate). These sterile swabs will be taken to the lab for aliquot culturing to yield 6 pitre dishes for each swab. The CFUs (colony forming units) from each pitre dish will be counted and analyzed at 48 and 72 hours. A comparison will be made using the cultures in Arm 1 and Arm 2 to determine if the parameters of the study has been met.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Class 1 clean (as defined by The American College of Surgeons)
* Hand and Feet extremities

Exclusion Criteria:

* Open wounds
* Pregnant
* Emergency surgeries
* Class 2-4 (as defined by The American College of Surgeons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Change in Time: Room to drape | Up to 60 minutes
  Minutes elapsed from patient ready for prep and ready for draping
Change in Time: ULTRAPREP bag use | Up to 60 minutes
  Minutes elapsed from ULTRAPREP placed on extremity to scrubbing complete
Colony forming units (CFU) Pre-Prep 48h | 48 hours after collection
  CFUs of bacteria per plate, collected upon arrival to pre-op area, measured after 48 hours growth
Colony forming units (CFU) Pre-Prep 72h | 72 hours after collection
  CFUs of bacteria per plate, collected upon arrival to pre-op area, measured after 72 hours growth
Colony forming units (CFU) Post-Prep 48h | 48 hours after collection
  CFUs of bacteria per plate, collected prior to draping, measured after 48 hours growth
Colony forming units (CFU) Post-Prep 72h | 72 hours after collection
  CFUs of bacteria per plate, collected prior to draping, measured after 72 hours growth

CONTACTS AND LOCATIONS:
Overall Officials: Pete Prados, Business, Study Director — PrepTech, LLC
Locations (1):
- PrepTech, LLC, Westlake, Louisiana, United States